CLINICAL TRIAL: NCT03598595
Title: A Phase 1/2 Study of Gemcitabine and Docetaxel in Combination With Hydroxychloroquine (Autophagy Inhibitor) in Patients With Recurrent Osteosarcoma
Brief Title: Gemcitabine, Docetaxel, and Hydroxychloroquine in Treating Participants With Recurrent or Refractory Osteosarcoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0224; NCI-2018-01414 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0224 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Recurrent Osteosarcoma; Refractory Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Docetaxel; Gemcitabine; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (hydroxychloroquine, gemcitabine, docetaxel) (Experimental): Participants receive hydroxychloroquine PO QD or BID on days 1-21, gemcitabine IV over 90 minutes on days 1 and 8, and docetaxel IV over 1 hours on day 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Docetaxel; Drug: Gemcitabine; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Drug: Hydroxychloroquine — Given PO

SUMMARY:
This phase I/II trial studies the side effects and best dose of hydroxychloroquine and how well it works when given together with gemcitabine and docetaxel in treating participants with osteosarcoma that has come back or does not respond to treatment. Drugs used in chemotherapy, such as gemcitabine, docetaxel, and hydroxychloroquine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and preliminary safety of hydroxychloroquine (HCQ) when administered with gemcitabine and docetaxel (G+D) in patients with recurrent/metastatic osteosarcoma. (Phase I) II. To determine whether gemcitabine and docetaxel (G+D) in combination with hydroxychloroquine (HCQ) increases the disease control rate in patients with recurrent/metastatic osteosarcoma at 4 months as compared to historic controls. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the objective response rate by Response Evaluation Criteria in Solid Tumors (RECIST) of the combination of G + D + HCQ in patients with recurrent/metastatic osteosarcoma.

II. To estimate the event-free survival (EFS), progression-free survival (PFS), and overall survival (OS) for patients with recurrent/metastatic osteosarcoma treated with G+D+HCQ.

III. To estimate the toxicity rates of oral HCQ when administered in conjunction with G+D.

IV. To investigate the pharmacokinetics (PK) of the combination in patients with recurrent/metastatic osteosarcoma.

EXPLORATORY OBJECTIVES:

I. To describe the metabolic response rates of G + D + HCQ in patients recurrent/metastatic measurable osteosarcoma by positron emission tomography (PET)/computed tomography (CT) at 6 weeks.

II. To assess pre-/post-treatment changes in autophagy biomarkers (autophagic vesicles, LC3B puncta, p62, and HMGB1), HSP27, and pHSP27 expression in tumor samples at baseline and during cycle #2 of treatment with G + D + HCQ.

III. To assess the relationship between probability of response and/or disease control and tumor HSP27, pHSP27, ALDH1A1, and HLTF expression.

IV. To complete functional proteomic profiling of autophagic and apoptotic pathways on tumor samples by RPPA and correlate findings with the probability response and disease control.

OUTLINE: This is a phase I, dose-escalation study of hydroxychloroquine followed by a phase II study.

Participants receive hydroxychloroquine orally (PO) once daily (QD) or twice daily (BID) on days 1-21, gemcitabine intravenously (IV) over 90 minutes on days 1 and 8, and docetaxel IV over 1 hours on day 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patient or patient's legally acceptable representative has provided informed consent
* Patients must have a pathological diagnosis of osteosarcoma at original diagnosis or time of recurrence
* Patients must have relapsed or become refractory to conventional therapy, with a regimen containing some combination of high dose methotrexate, doxorubicin, cisplatin, and/or ifosfamide
* Patients may have either unresectable or potentially resectable disease. However, patients with potentially resectable disease must be willing to await surgery until after the primary efficacy endpoint is reached at 4 months
* Patients must have measurable disease by RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2. Use Karnofsky for patients > 16 years old and Lansky for patients =< 16
* Has archived tumor tissue and is willing to provide a tumor block or unstained slides or the patient is willing to undergo a pretreatment biopsy. Biopsy during cycle #2 of therapy is required. Biopsy at progression is strongly encouraged but will be optional
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L
* Platelet count >= 100 x 10^9/L
* Hemoglobin > 8 g/dL
* Prothrombin time (PT) or partial thromboplastin time (PTT) < 1.5 x upper limit of normal (ULN), except subjects on anticoagulation for venous thromboembolism
* Calculated creatinine clearance or radioisotope glomerular filtration rate (GFR) > 60 mL/min
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 x ULN for age
* Total bilirubin < 1.5 x ULN for age
* Serum albumin >= 2

Exclusion Criteria:

* Any disorder that compromises the ability of the patient or patient's legally acceptable representative to give written informed consent and/or to comply with the study procedures
* Patients who will not be available for protocol required study visits, to the best of the subject and investigator's knowledge
* History of hypersensitivity to any of the study agents (gemcitabine, docetaxel, or hydroxychloroquine) or to any component of the formulation
* Patients who have previously received gemcitabine or docetaxel
* Men and woman of reproductive potential, unwilling to practice a highly effective method of birth control for the duration of the study and continuing for 2 weeks (for women) and 12 weeks (for men) after receiving the last dose of study drug. Highly effective methods of birth control include sexual abstinence (men, women); vasectomy or a condom used with spermicide (men) in combination with barrier methods, hormonal birth control or intrauterine device (IUD) (women)
* Women who are lactating/breastfeeding or planning to become pregnant during the duration of the study
* History or current diagnosis of a second neoplasm. Exception: adequately treated non-melanoma skin cancer, curatively treated in-situ disease, or other solid tumors curatively treated with no evidence of disease for >= 2 years
* Myocardial infarction within 6 months of study day 1, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina, or unstable cardiac arrhythmia requiring medication, or uncontrolled hypertension (systolic > 160 mmHg or diastolic > 100 mmHg)
* Active infection requiring intravenous (IV) antibiotics within 2 weeks of study enrollment
* Significant gastrointestinal disorder(s) that in the opinion of the investigator (e.g., Crohn's disease, ulcerative colitis, extensive gastrointestinal resection) may influence drug absorption
* Known positive test for human immunodeficiency virus (HIV)
* Subjects with acute hepatitis B and C are not eligible. Subjects with chronic hepatitis B or C are eligible if their condition is stable and, in the opinion of the investigator and Amgen physician, if consulted, would not pose a risk to subject safety
* Toxicities from prior anti-tumor therapy not resolved to Common Terminology Criteria for Adverse Events (CTCAE) grade 0 or 1, or to levels dictated in the eligibility criteria. Grade 2 toxicities from prior anti-tumor therapy that are considered irreversible (defined as having been present and stable for > 4 weeks), such as stable grade 2 peripheral neuropathy or ifosfamide-related proteinuria, may be allowed if they are not otherwise described in the exclusion criteria AND there is agreement to allow by the principal investigator
* Prior participation in an investigational study and/or procedure within 21 days of study day 1
* Anti-tumor therapy within 21 days of study day 1 including chemotherapy, antibody therapy, or other investigational agent. Enrollment of subjects that have received molecularly targeted agents less than 28 days prior to study day 1 will be permitted if more than 14 days and at least 5 drug half-lives have passed prior to receiving the first dose of HCQ
* Major surgery within 28 days of study day 1
* Any co-morbid medical disorder that may increase the risk of toxicity, in the opinion of the investigator
* All herbal supplements, vitamins, and nutritional supplements taken within the last 30 days prior to dosing on day 1 (and continued use, if appropriate), must be reviewed and approved by the principal investigator (PI)
* Patients with pre-existing maculopathy or retinopathy of the eye

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of hydroxychloroquine (Phase I) | Up to 21 days
Disease control rate (Phase II) | At 4 months

SECONDARY OUTCOMES:
Event free survival | From enrollment to disease progression, death, or discontinuation of treatment for any reason, assessed up to 2 years
Overall response (complete response [CR] or partial response [PR] versus not CR or PR) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John A Livingston, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org